CLINICAL TRIAL: NCT00006385
Title: Phase II Evaluation of Immunization With an HLA-A2 Multi-Epitope Peptide Vaccine Containing MART-1 (NSC #672643), gp100 (NSC #683472), and Tyrosinase (NSC #699048) Peptides Alone or in Combination With GM-CSF, IFN Alpha-2b, or GM-CSF + IFN Alpha-2b in Patients With Metastatic Melanoma
Brief Title: Vaccine Therapy With or Without Biological Therapy in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068263; E-1696
Record Dates: First submitted 2000-10-04; First posted 2003-01-27 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2002-12

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — MART-1 Antigen; incomplete Freund's adjuvant; Interferon-alpha; sargramostim

INTERVENTIONS:
Biological: MART-1 antigen
Biological: gp100 antigen
Biological: incomplete Freund's adjuvant
Biological: recombinant interferon alfa
Biological: sargramostim
Biological: tyrosinase peptide

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Biological therapies such as sargramostim and interferon alfa use different ways to stimulate the immune system and stop cancer cells from growing. It is not yet known if vaccine therapy if more effective with or without biological therapy for melanoma.

PURPOSE: Randomized phase II trial to compare the effectiveness of vaccine therapy with or without biological therapy in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine immune response of vaccination with melanoma associated antigens (MART-1:27-35, gp100:209-217 (210M), and tyrosinase:368-376 (370D)) on the number of peptide specific CD8+ T-cell precursors in HLA-A2 positive patients with metastatic melanoma.
* Determine the influence of sargramostim (GM-CSF) and/or interferon alfa-2b (IFN-A) on the immune responses of these patients and toxicity of this melanoma peptide vaccine.
* Determine any antitumor and anti-pigmentary response that may result from immunization against MART-1, gp100 and tyrosinase peptides, and determine the relationship between such clinical observations and immune responses against lineage antigens with or without GM-CSF and/or IFN-A.
* Compare the relapse free survival and overall survival of patients treated with melanoma peptide vaccine alone or in combination with GM-CSF and/or IFN-A.

OUTLINE: This is a randomized, multicenter study.

Patients are randomized to 1 of 4 treatment arms.

* Arm I: Patients receive multiepitope peptide (MEP) vaccine comprising MART-1:27-35, gp100:209-217 (210M), and tyrosinase:368-376 (370D) peptides. Each peptide is separately emulsified in Montanide ISA-51 and administered subcutaneously (SC) (for a total of 2 injections per peptide) on days 1 and 15.
* Arm II: Patients receive MEP vaccine as in arm I and sargramostim (GM-CSF) subcutaneously (SC) daily on days 1-14.
* Arm III: Patients receive MEP vaccine as in arm I and interferon alfa-2b SC three times a week.
* Arm IV: Patients receive MEP vaccine as in arm I, GM-CSF as in arm II, and interferon alfa-2b as in arm III.

Treatment continues every 4 weeks for a maximum of 13 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 92 patients (23 per arm) will be accrued for this study within 13-16 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage IV melanoma
* Measurable disease

  * At least 1 lesion must be a minimum of 1.0 cm in diameter
  * Bone metastases are not considered to be measurable disease
  * No prior radiotherapy to area of measurable disease unless there is clearly progressive disease in this site or measurable disease exists outside the area of prior radiotherapy
* HLA-A2 positive
* No brain disease by MRI or CT scan within 4 weeks prior to randomization

  * Prior brain disease allowed if no evidence of active disease by 2 successive MRI evaluations completed at least 3 months apart

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* WBC at least 4,000/mm^3
* Platelet count at least 100,000/mm^3
* Lymphocyte count greater than 700/mm ^3

Hepatic:

* SGOT no greater than 2 times upper limit of normal (ULN)
* Bilirubin no greater than 2 times ULN
* Alkaline phosphatase and lactic dehydrogenase no greater than 2 times ULN

Renal:

* Creatinine no greater than 1.8 mg/dL

Other:

* No significant detectable infection
* HIV negative
* No other malignancy within the past 5 years except:

  * Any carcinoma in situ
  * Lobular carcinoma in situ of the breast
  * Carcinoma in situ of the cervix
  * Atypical melanocytic hyperplasia
  * Melanoma in situ
  * Basal cell or squamous cell skin cancer
* No autoimmune disorders or conditions of immunosuppression
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior MART-1:27-35, gp100:209-217 (210M), or tyrosinase:368-376 (370D) peptide
* Greater than 4 weeks since prior adjuvant immunotherapy, including sargramostim (GM-CSF) or interferon alfa-2b

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)

Endocrine therapy:

* At least 2 weeks since prior and no concurrent systemic corticosteroids, including oral steroids (i.e., prednisone, dexamethasone); continuous use of topical steroid creams or ointments; or any inhalers containing steroids

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy for local control or palliation and recovered

Surgery:

* Recovered from any prior major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-09; Primary Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M. Kirkwood, MD, Study Chair — University of Pittsburgh
Locations (32):
- United States (32):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Tuft-New England Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - Scott and White Hospital, Temple, Texas
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
  - Veterans Affairs Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin

REFERENCES:
- [Result] Schaefer C, Butterfield LH, Lee S, Kim GG, Visus C, Albers A, Kirkwood JM, Whiteside TL. Function but not phenotype of melanoma peptide-specific CD8(+) T cells correlate with survival in a multiepitope peptide vaccine trial (ECOG 1696). Int J Cancer. 2012 Aug 15;131(4):874-84. doi: 10.1002/ijc.26481. Epub 2012 Jan 11. PMID 22021080
- [Result] Kirkwood JM, Lee S, Moschos SJ, Albertini MR, Michalak JC, Sander C, Whiteside T, Butterfield LH, Weiner L. Immunogenicity and antitumor effects of vaccination with peptide vaccine+/-granulocyte-monocyte colony-stimulating factor and/or IFN-alpha2b in advanced metastatic melanoma: Eastern Cooperative Oncology Group Phase II Trial E1696. Clin Cancer Res. 2009 Feb 15;15(4):1443-51. doi: 10.1158/1078-0432.CCR-08-1231. PMID 19228745
- [Result] Kirkwood JM, Lee S, Land S, et al.: E1696: final analysis of the clinical and immunological results of a multicenter ECOG phase II trial of multi-epitope peptide vaccination for stage IV melanoma with MART-1 (27-35), gp100 (209-217, 210M), and tyrosinase (368-376, 370D) (MGT) +/- IFNα2b and GM-CSF. [Abstract] J Clin Oncol 22 (Suppl 14): A-7502, 710s, 2004.
- [Result] Kirkwood JM, Lee S, Land S, et al.: E1696: phase II trial of multi-epitope peptide vaccination for melanoma with MGT (MART-1 (27-35), gp100 (209-217, 210M) and tyrosinase (368-376, 370D))+/- IFN alfa-2b and GM-CSF--immunological and clinical results. [Abstract] 22: A-2850, 709, 2003.